CLINICAL TRIAL: NCT06778213
Title: A Randomized Placebo-controlled Double-blind Clinical Study for Evaluation of the Efficacy of Allergen-specific Immunotherapy Using Clinical and Biomarker Assessment in an Allergen Exposure Chamber and During Natural Exposure in Patients With House Dust Mite-triggered Allergic Rhinoconjunctivitis RANSES
Brief Title: Evaluation of the Efficacy of Allergen-specific Immunotherapy Using Assessment in an Allergen Exposure chamber-a Randomized Placebo-controlled Double-blind Study
Acronym: RANSES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Collaborators: ALL-MED Medical Research Institute, Wroclaw, Poland (Unknown); Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Marek Jutel, professor, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALL-MED
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: allergen-specific immunotherapy; biomarker assessment; allergen exposure chamber; house dust mite; allergic rhinoconjunctivitis

STUDY DESIGN:
Intervention Model Description: A randomized placebo-controlled double-blind study
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- verum (Active Comparator): Immunotherapy - NovoHelisen Depot according to desensitisation protocol 5 times weekly increasing injections 250-5000 TU, 10 times monthly maintenance injections 5000 TU
  Interventions: Biological: NovoHelisen Depot
- placebo (Placebo Comparator): 5 times weekly increasing placebo injections, 10 times monthly placebo injections
  Interventions: Biological: NovoHelisen Depot

INTERVENTIONS:
Biological: NovoHelisen Depot — allergen immunotherapy treatment for 12 months with house dust mite allergen preparation

SUMMARY:
The main objective of the study is to measure and correlate clinical parameters suitable for the assessment of allergen immunotherapy (AIT) with an aluminum hydroxide-adsorbed preparation of house dust mite (Dermatophagoides pteronyssinus/ Dermatophagoides farinae) allergens in adults with moderate to severe allergic rhinitis/rhinoconjunctivitis with or without controlled allergic bronchial asthma caused by house dust mite (HDM) allergens. The assessment of clinical responses will be evaluated following an allergen challenge in allergen exposure chamber (AEC) before and during the course of AIT. Patients' response to therapy will be evaluated as well as in the AEC and by patient's personal environment (Diary).

DETAILED DESCRIPTION:
This clinical trial will be performed as a randomized, double-blind, placebo-controlled phase IV study in adult patients. Thus, 2 parallel groups, one active treated and one placebo group, will be investigated. Patients from 18 to 65 years of age with moderate to severe allergic rhinitis or rhinoconjunctivitis to HDM allergens, with or without controlled allergic bronchial asthma, will be enrolled.

The efficacy will be evaluated using an AEC (TNSS) and additionally in the patient's natural environment (SMS). The screening phase will begin approximately in May and last until September 2024. All patients fulfilling the eligibility criteria at Screening Visit 1 (S1) will perform an AEC visit (AEC-pre) in October, followed by an e-Diary phase in November, December (Diary-pre). For the assessment of the pre-treatment score 4 consecutive weeks will be recorded and at least 2 consecutive weeks with complete daily entries must available. Adequate symptoms are defined as patient randomization criteria in the respective section of the synopsis/protocol. After randomization, patients will be treated for approximately 10 months. Afterwards a second Diary phase (Diary-post) will be performed. For the assessment of the post-treatment score, at least 2 consecutive weeks with complete daily entries must be available. Then, a second, posttreatment challenge (AEC-post) will follow. Last patient last visit is planned for January 2026. For the trial approximately 80 male and female outpatients (18 to 65 years of age) will be screened, and 67 patients will be randomized 1:1 verum/placebo. It is assumed, that this number of patients will yield a total of at least 60 patients with available post-treatment assessments, assuming a dropout rate of 10%. Additionally, data from 11 healthy subjects from a previous study with an identical setting will be included in the correlation analysis. There will be no replacement strategy employed for patients dropping out prematurely.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for trial participation, patients must meet all the following inclusion criteria:

1. Written informed consent given from patient according to local requirements before any trial-related activities started (a trial-related activity is any procedure that would not have been performed during the routine management of the patient)
2. Legally competent male or female outpatient between 18 and ≤ 65 years
3. IgE-mediated moderate to severe allergic rhinitis or rhinoconjunctivitis with or without allergic asthma caused by HDM allergens documented by

   Positive Skin prick test (SPT) result to D. pteronyssinus allergens:

   D. pteronyssinus test solution (wheal diameter) ≥ 3 mm and Positive histamine-control reaction (wheal diameter) ≥ 3 mm and Negative NaCl-control reaction (wheal diameter) < 2 mm Immunoassay result for specific IgE ≥ 0.70 kU/L to D. pteronyssinus
4. Symptoms of rhinitis or rhinoconjunctivitis e.g., during the months October to February or over the entire year for at least 2 years before enrolment.
5. Assessment of persistent, moderate-severe rhinitis acc. to ARIA guidelines (Brozek et al.

2017, Bousquet et al. 2001) Symptoms for 4 or more consecutive weeks in the previous years and for at least 4 days per week during those weeks More than one of the symptoms evaluated as "troublesome" by the patients and/or impairing their daily activities, leisure or sport, school, or work and/or involving sleep disturbance 6. Symptoms requiring regular intake of anti-symptomatic medication 7. Previous symptomatic anti-allergic medication for at least 2 seasons prior to enrolment 8. At entry to this trial: No diagnosis of bronchial asthma in medical history or confirmed diagnosis of asthma as being "well controlled" according to GINA recommendation (GINA 2022)

Exclusion Criteria:

General criteria:

1. Patients are unable to understand and comply with the requirements of the trial, as judged by the investigator
2. Currently participating in another clinical trial or participating in any other clinical trial within 30 days prior informed consent for this trial
3. Low adherence to trial procedures expected or inability to understand instructions/trial documents
4. Involvement in the planning and conduct of the trial
5. Any relationship of dependence with the investigator
6. Previous randomization to treatment in the present trial
7. Mentally disabled
8. Institutionalized due to an official or judicial order For female patients with childbearing potential (i.e., females who are not chemically or surgically sterilized or females who are not post-menopausal)
9. Positive urine pregnancy test or pregnant
10. Wish to become pregnant during the course of the trial
11. Not using highly effective and reliable contraception, as judged by the investigator (reliable and highly effective methods of birth control defined as a failure rate of less than 1% per year [CTFG recommendations 2020]) during the trial. Sexual abstinence is an allowed method of birth control (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.) Males are not required to use any contraception during the study.
12. Wish to breastfeed or breastfeeding

    Immunotherapy criteria:
13. History of a confirmed anaphylaxis after an AIT injection
14. Current treatment with any kind of AIT
15. AIT with HDM allergoids or allergens within the last 5 years
16. AIT with unknown allergen within the last 5 years Sensitization criteria
17. Clinically relevant symptoms to perennial and seasonal allergens which interfere with the assessment period of October to January. Exceptions are symptoms to allergens of cat and dog, if the patient has no direct contact to these animals.

    Diseases and health status:
18. Clinically relevant chronic rhinoconjunctival or respiratory symptoms related to other reasons than allergy
19. Chronic persistent rhinitis symptoms for 20 years or longer
20. Forced expiratory volume in 1 second (FEV1) < 70 % of predicted normal values according to Quanjer (Quanjer et al. 2012) under adequate asthma treatment according to GINA recommendation (GINA 2022)
21. Uncontrolled or partly controlled asthma according to GINA recommendation (GINA 2022)
22. Asthma exacerbation within the last 6 months prior to randomization defined as unscheduled doctors visit, hospitalization, or emergency unit visit requiring the use of systemic corticosteroids or change of controller medication
23. Severe acute or chronic diseases (e.g., COVID-19, chronic urticaria, mastocytosis, active tuberculosis, diabetes mellitus type I, malignant neoplasia, chronic renal failure), severe inflammatory diseases (liver, kidneys)
24. Autoimmune diseases, immune defects including immunosuppression, immune-complexinduced immunopathies (e.g., HIV, post-transplant patients, lupus erythematodes [SLE], vitiligo, Grave's disease, multiple sclerosis)
25. Severe psychiatric and psychological disorders including impairment of cooperation (e.g., alcohol or drug abuse)
26. Recurrent seizures (e.g., febrile convulsion, untreated epilepsy)
27. Irreversible secondary alterations of the reactive organ (e.g., emphysema, bronchiectasis)
28. For assessment the normal reference ranges of the central laboratory should be applied. If out of range, laboratory values greater than grade 1 according to the FDA Guidance for Industry (Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials) will lead to exclusion of the patient.

    Medications:
29. Use of β-blockers (locally or systemically) and/or angiotensin-converting enzyme (ACE) inhibitors
30. Contraindication for use of adrenalin (e.g., acute, or chronic symptomatic coronary heart disease, severe hypertension)
31. Completion or ongoing treatment with anti-IgE-antibodies (e.g., omalizumab) or anti IL4/IL13 antibodies (e.g., dupilumab) or other biological medication interfering with the TH2 pathway
32. Completed or ongoing long-term treatment with tranquilizer or other psychoactive drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Total nasal symptom score | 12 months
  The primary efficacy analysis is the analysis of correlation between TNSS recorded in the AEC and the average CSMS over 2 weeks as recorded in the eDiary.

SECONDARY OUTCOMES:
Change of the TNSS | 12 months
  Change of the TNSS at 120 minutes recorded in the AEC from pre-treatment to post treatment, calculated as post treatment TNSS - pre-treatment TNSS, and Change in average CSMS from pre-treatment to post-treatment calculated as post treatment CSMS - pre-treatment CSMS
Change in average CSMS | 12 months
  Change in average CSMS from pre-treatment to post-treatment calculated as post treatment CSMS - pre-treatment CSMS

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka M Chuda, MSc, Study Director — ALL-MED Specjalistyczna Opieka Medyczna. Medyczny Instytut Badawczy
Locations (1):
- ALL-MED Medical Research Institute, Wroclaw, DL, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zemelka-Wiacek M, Kosowska A, Winiarska E, Sobanska E, Jutel M. Validated allergen exposure chamber is plausible tool for the assessment of house dust mite-triggered allergic rhinitis. Allergy. 2023 Jan;78(1):168-177. doi: 10.1111/all.15485. Epub 2022 Sep 1. PMID 35980665
- [Background] Kosowska A, Zemelka-Wiacek M, Smolinska S, Wyrodek E, Adamczak B, Jutel M. Clinical validation of grass pollen exposure chamber in patients with allergic rhinitis triggered by timothy grass. Clin Exp Allergy. 2024 Jul;54(7):489-499. doi: 10.1111/cea.14482. Epub 2024 Apr 14. PMID 38616622
- [Background] Jutel M, Zemelka-Wiacek M, Okamoto Y, Pfaar O. Algorithms in Allergy: Assessment of Rhinitis Using Allergen Exposure Chambers. Allergy. 2025 Mar;80(3):904-907. doi: 10.1111/all.16444. Epub 2024 Dec 17. No abstract available. PMID 39688144
- [Background] Zemelka-Wiacek M, Kosowska A, Jutel M. Symptom Assessment of Patients with Allergic Rhinitis Using an Allergen Exposure Chamber. J Vis Exp. 2023 Mar 3;(193). doi: 10.3791/64801. PMID 36939263
- See also: ALLEC Allergen Exposure Chamber — https://www.all-med.wroclaw.pl/allec_chamber_facility.html